CLINICAL TRIAL: NCT01095445
Title: EXtended Therapy in Genotype 3 Infected Patients Who do Not AChieve a Treatment Response at Week 4 (RVR) But do Achieve a Complete Early Virologic Response (cEVR)
Brief Title: EXtended Therapy in Hepatitis C Genotype 3 Infected Patients
Acronym: EXACT-R(3)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unlikely to recruit the adequate number of patients within a reasonable timeline
Sponsor: University Health Network, Toronto (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXACT-R(3)
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Hepatitis C
Keywords: hepatitis C; genotype 3; end of treatment response; relapse rate; rapid virologic response; complete early virologic response
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care treatment (No Intervention): Participants will be randomized to receive only the standard 24 weeks of therapy (Peginterferon alfa-2b plus ribavirin).
- Extended therapy (Active Comparator): Participants will be randomized to receive 24 weeks of therapy (Peginterferon alfa-2b plus ribavirin) in addition to their standard of care therapy.
  Interventions: Drug: Peginterferon alfa-2b (Pegetron) plus ribavirin (Rebetol)

INTERVENTIONS:
Drug: Peginterferon alfa-2b (Pegetron) plus ribavirin (Rebetol) — Dosage Form: Pegetron - powder for solution; Rebetol - capsules Strength: Pegetron Redipen - 120 mcg per pen; Rebetol - 200 mg Route of Administration: Pegetron - subcutaneous; Rebetol - oral
  Other Names: Pegetron; Rebetol
  Arms: Extended therapy

SUMMARY:
The purpose of this study is to evaluate the effect of 48 vs 24 weeks of treatment with Peginterferon alfa-2b plus weight-based ribavirin on Sustained Virologic Response (SVR) and relapse rates in patients infected with genotype 3 chronic hepatitis C (CHC) who do not achieve a Rapid Virologic Response (RVR) but attain a complete Early Virologic Response (cEVR).

DETAILED DESCRIPTION:
This study plans to address the issue of whether increasing the duration of therapy from 24 weeks to 48 weeks with PegIFNα2b 1.5mg/kg/week and using weight-based ribavirin (15mg/kg) may reduce relapse rates and thereby increase SVR rates in patients infected with genotype 3 who fail to achieve an RVR but do achieve a complete cEVR defined as undetectable HCV RNA (ie. <50 or <15 IU/ml by 12 weeks). This study is necessary because although most patients with genotype 3 ultimately become HCV RNA undetectable during treatment, relapse after discontinuation of therapy remains a major cause of failure to achieve SVR. This is a very important issue given that to date none of the new small molecule drugs appear effective against genotype 3 meaning that at the present time patients with genotype 3 infection have no other options. Relapse is particularly common in patients with advanced liver disease but it has been shown that if SVR can be achieved in patients with advanced disease, the risk of liver failure is significantly reduced, as may be the risk of hepatocellular carcinoma (HCC). As a consequence the need for liver transplantation is diminished and survival is improved. Identifying strategies to reduce relapse and improve rates of SVR are therefore critical.

Certain individuals are at greater risk of infection with genotype 3. In the Western world, the main risk groups are current or former drug users (IDU) and immigrants raised in South Asia (India and Pakistan) where infection likely occurs early in childhood due to exposure to contaminated instruments, needles, etc.

A second potential benefit of achieving SVR is reduction in the rate of diabetes. Diabetes has been demonstrated to be more common in those infected with Hepatitis C than in the general population - this observation was made by examination of the NHANES population based database. The prelude to the development of Type 2 diabetes is insulin resistance. Insulin resistance (IR) is present in about one third of patients chronically infected with HCV - the rate being highest in those with cirrhosis and in those who are overweight or obese. Early data indicates that although the presence of insulin resistance impairs interferon responsiveness if SVR can be achieved, insulin resistance is lost. Studies of IR in individuals infected with genotype 3 HCV are lacking. Independent of HCV infection, being born South Asian is a risk factor for Type 2 diabetes.

The issue of insulin resistance and the effectiveness of antiviral therapy in chronic hepatitis C has been addressed exclusively in Caucasians infected with genotype 1. Recent data from Japan indicates that in patients with diabetes and hepatitis C successful eradication of HCV RNA may simultaneously prevent subsequent diabetes and presumably the systemic complications of this disease.

There is little data on the rate of RVR in the South Asian population as few therapeutic trials in patients with genotype 3 infections have been reported from Pakistan and India. Estimates can only be obtained from studies performed in Caucasians from Northern Europe and North America. In the trial by Shiffman the rate of RVR in those with genotype 3 infection was 62% and preliminary report from the trial of Albuferon in those with genotype 2 and 3 indicate RVR rates ranged from 44-60% in Asians -this figure included all Asians.

There are several reasons to specifically address ways to improve the outcome of antiviral therapy in patients infected with genotype 3 CHC. Firstly virtually all treatment studies report on a combined rate of SVR achieved in genotypes 2 and 3 even though the evidence has suggested that the response to therapy is different between these two genotypes. Within populations of patients with genotype 3 infection, there may be differences as well. South Asians are predominantly infected with genotype 3a, while injection drug users typically have genotype 3b infection. There are no formal trials published in the English literature of antiviral therapy in South Asians or comparing subtypes of genotype 3.

In patients infected with genotype 1 slow response to antiviral therapy i.e. lack of RVR, is associated with a significantly higher rate of relapse in those who go on to achieve undetectable HCV RNA at 12 weeks rather than at 4 weeks into treatment. Extending treatment for a further six months reduces this relapse rate considerably. By extending treatment in patients infected with genotype 3 who had previously relapsed following only 14 weeks of therapy to 24 weeks reduced relapse rates. Thus, it is anticipated that by extending treatment from 24 to 48 weeks in those who fail to achieve a RVR (i.e. slow responders) but who do achieve a complete EVR we hope to prevent relapse off treatment. A potential added benefit of achieving SVR in this patient population, many of whom are already at high risk of T2DM, is that it may reduce the virally mediated component of IR.

ELIGIBILITY:
Inclusion Criteria:

* Infected with only genotype 3, hepatitis C
* Treatment naïve before current course of therapy
* A positive HCV RNA test result at Week 4 (no RVR)
* A negative HCV RNA test result at Week 12 (cEVR)
* A recent liver biopsy (within 3 years prior to study entry) is required. If the patient has either liver biopsy proven cirrhosis in the past or has splenomegaly with features of cirrhosis on ultrasound and/or thrombocytopenia (<150x109/ml) at any time in the past or has a Fibroscan reading of 10 or above or has a Fibrotest score of 0.75 or above (equivalent to F3 on the METAVIR scale), a biopsy will not be required. A copy of the latest report must be available.

Exclusion Criteria:

* Under age 18
* Co-infection with HIV or Hepatitis B or any other HCV genotype in addition to genotype 3
* Prior treatment for Hepatitis C aside from herbal remedies
* Evidence of decompensated liver disease, such as ascites, bleeding varices, hepatic encephalopathy or jaundice (conjugated hyperbilirubinemia)
* INR > 1.3 at baseline
* Platelet count <70 X 109/μl at baseline
* Those subjects with diabetes and/or systemic hypertension will need to have ocular examinations (as per standard of care [SOC]) prior to treatment and will be excluded if they are found to have a diabetic retinopathy, optic nerve disorders, retinal hemorrhage or any other clinically significant abnormality
* Pre-existing psychiatric conditions including:

  * Current moderate or severe depression despite appropriate therapy.
  * Active suicidal ideation or previous attempt at suicide
  * Patients with a history of severe psychiatric disorder (may be included if so desired by the investigator but pretreatment psychiatric evaluation is required (SOC)).
  * Clinical diagnosis of current substance abuse: Alcohol (>40g/d), injection drugs, inhalational drugs (not including marijuana), psychotropics, narcotics, cocaine use, prescription or over the counter drugs within one year of the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
End of treatment response | 24 weeks following end of therapy
  Undetectable hepatitis C virus (HCV) RNA at 24 weeks following end of therapy

SECONDARY OUTCOMES:
Relapse rate | 24 weeks following end of therapy
  Undetectable HCV RNA at end of treatment but detectable HCV RNA at 24 weeks following end of therapy

CONTACTS AND LOCATIONS:
Overall Officials: E. Jenny Heathcote, MB,BS,MD,FRCP,FRCP(C), Principal Investigator — University Health Network - Toronto Western Hospital
Locations (12):
- Canada (12):
  - Calgary Heart Centre, Calgary, Alberta
  - Hys Med Centre, Edmonton, Alberta
  - Liver and Intestinal Research Centre, Vancouver, British Columbia
  - Dr. John D Farley Medical Office, Vancouver, British Columbia
  - Pacific Gastroenterology Assoc, Vancouver, British Columbia
  - Hotel Dieu Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Dr. Dalia El-Ashry clinic, Mississauga, Ontario
  - Credit Valley Med Arts Centre, Mississauga, Ontario
  - Toronto General Hospital - Dr. M. Sherman, Toronto, Ontario
  - Toronto Western Hospital - Liver Clinic, Toronto, Ontario
  - SMBD Jewish Gen Hosp, Montreal, Quebec

REFERENCES:
- [Background] Hadziyannis SJ, Sette H Jr, Morgan TR, Balan V, Diago M, Marcellin P, Ramadori G, Bodenheimer H Jr, Bernstein D, Rizzetto M, Zeuzem S, Pockros PJ, Lin A, Ackrill AM; PEGASYS International Study Group. Peginterferon-alpha2a and ribavirin combination therapy in chronic hepatitis C: a randomized study of treatment duration and ribavirin dose. Ann Intern Med. 2004 Mar 2;140(5):346-55. doi: 10.7326/0003-4819-140-5-200403020-00010. PMID 14996676
- [Background] Zeuzem S, Hultcrantz R, Bourliere M, Goeser T, Marcellin P, Sanchez-Tapias J, Sarrazin C, Harvey J, Brass C, Albrecht J. Peginterferon alfa-2b plus ribavirin for treatment of chronic hepatitis C in previously untreated patients infected with HCV genotypes 2 or 3. J Hepatol. 2004 Jun;40(6):993-9. doi: 10.1016/j.jhep.2004.02.007. PMID 15158341
- [Background] Powis J, Peltekian KM, Lee SS, Sherman M, Bain VG, Cooper C, Krajden M, Deschenes M, Balshaw RF, Heathcote EJ, Yoshida EM; Canadian Pegasys Study Group. Exploring differences in response to treatment with peginterferon alpha 2a (40kD) and ribavirin in chronic hepatitis C between genotypes 2 and 3. J Viral Hepat. 2008 Jan;15(1):52-7. doi: 10.1111/j.1365-2893.2007.00889.x. PMID 18088245
- [Background] Dalgard O, Bjoro K, Hellum KB, Myrvang B, Ritland S, Skaug K, Raknerud N, Bell H. Treatment with pegylated interferon and ribavarin in HCV infection with genotype 2 or 3 for 14 weeks: a pilot study. Hepatology. 2004 Dec;40(6):1260-5. doi: 10.1002/hep.20467. PMID 15558712
- [Background] Lagging M, Langeland N, Pedersen C, Farkkila M, Buhl MR, Morch K, Dhillon AP, Alsio A, Hellstrand K, Westin J, Norkrans G; NORDynamIC Study Group. Randomized comparison of 12 or 24 weeks of peginterferon alpha-2a and ribavirin in chronic hepatitis C virus genotype 2/3 infection. Hepatology. 2008 Jun;47(6):1837-45. doi: 10.1002/hep.22253. PMID 18454508
- [Background] Mangia A, Santoro R, Minerva N, Ricci GL, Carretta V, Persico M, Vinelli F, Scotto G, Bacca D, Annese M, Romano M, Zechini F, Sogari F, Spirito F, Andriulli A. Peginterferon alfa-2b and ribavirin for 12 vs. 24 weeks in HCV genotype 2 or 3. N Engl J Med. 2005 Jun 23;352(25):2609-17. doi: 10.1056/NEJMoa042608. PMID 15972867
- [Background] Dalgard O, Bjoro K, Ring-Larsen H, Bjornsson E, Holberg-Petersen M, Skovlund E, Reichard O, Myrvang B, Sundelof B, Ritland S, Hellum K, Fryden A, Florholmen J, Verbaan H; North-C Group. Pegylated interferon alfa and ribavirin for 14 versus 24 weeks in patients with hepatitis C virus genotype 2 or 3 and rapid virological response. Hepatology. 2008 Jan;47(1):35-42. doi: 10.1002/hep.21975. PMID 17975791
- [Background] Shiffman ML, Suter F, Bacon BR, Nelson D, Harley H, Sola R, Shafran SD, Barange K, Lin A, Soman A, Zeuzem S; ACCELERATE Investigators. Peginterferon alfa-2a and ribavirin for 16 or 24 weeks in HCV genotype 2 or 3. N Engl J Med. 2007 Jul 12;357(2):124-34. doi: 10.1056/NEJMoa066403. PMID 17625124
- [Background] Bain VG, Kaita KD, Marotta P, Yoshida EM, Swain MG, Bailey RJ, Patel K, Cronin PW, Pulkstenis E, McHutchison JG, Subramanian GM. Safety and antiviral activity of albinterferon alfa-2b dosed every four weeks in genotype 2/3 chronic hepatitis C patients. Clin Gastroenterol Hepatol. 2008 Jun;6(6):701-6. doi: 10.1016/j.cgh.2008.02.056. Epub 2008 May 7. PMID 18467185
- [Background] Vigani AG, Pavan MH, Tozzo R, Goncales ES, Feltrin A, Fais VC, Lazarini MS, Goncales NS, Goncales FL Jr. Comparative study of patients with chronic hepatitis C virus infection due to genotypes 1 and 3 referred for treatment in southeast Brazil. BMC Infect Dis. 2008 Dec 4;8:164. doi: 10.1186/1471-2334-8-164. PMID 19055835
- [Background] Mangia A, Minerva N, Bacca D, Cozzolongo R, Agostinacchio E, Sogari F, Scotto G, Vinelli F, Ricci GL, Romano M, Carretta V, Petruzzellis D, Andriulli A. Determinants of relapse after a short (12 weeks) course of antiviral therapy and re-treatment efficacy of a prolonged course in patients with chronic hepatitis C virus genotype 2 or 3 infection. Hepatology. 2009 Feb;49(2):358-63. doi: 10.1002/hep.22679. PMID 19072829
- [Background] Farooqi JI, Farooqi RJ. Conventional interferon alfa-2b and ribavirin for 12 versus 24 weeks in HCV genotype 2 or 3. J Coll Physicians Surg Pak. 2008 Oct;18(10):620-4. doi: 10.2008/JCPSP.620624. PMID 18940119
- [Background] von Wagner M, Huber M, Berg T, Hinrichsen H, Rasenack J, Heintges T, Bergk A, Bernsmeier C, Haussinger D, Herrmann E, Zeuzem S. Peginterferon-alpha-2a (40KD) and ribavirin for 16 or 24 weeks in patients with genotype 2 or 3 chronic hepatitis C. Gastroenterology. 2005 Aug;129(2):522-7. doi: 10.1016/j.gastro.2005.05.008. PMID 16083709
- [Background] Veldt BJ, Heathcote EJ, Wedemeyer H, Reichen J, Hofmann WP, Zeuzem S, Manns MP, Hansen BE, Schalm SW, Janssen HL. Sustained virologic response and clinical outcomes in patients with chronic hepatitis C and advanced fibrosis. Ann Intern Med. 2007 Nov 20;147(10):677-84. doi: 10.7326/0003-4819-147-10-200711200-00003. PMID 18025443
- [Background] Mehta SH, Brancati FL, Strathdee SA, Pankow JS, Netski D, Coresh J, Szklo M, Thomas DL. Hepatitis C virus infection and incident type 2 diabetes. Hepatology. 2003 Jul;38(1):50-6. doi: 10.1053/jhep.2003.50291. PMID 12829986
- [Background] Moucari R, Asselah T, Cazals-Hatem D, Voitot H, Boyer N, Ripault MP, Sobesky R, Martinot-Peignoux M, Maylin S, Nicolas-Chanoine MH, Paradis V, Vidaud M, Valla D, Bedossa P, Marcellin P. Insulin resistance in chronic hepatitis C: association with genotypes 1 and 4, serum HCV RNA level, and liver fibrosis. Gastroenterology. 2008 Feb;134(2):416-23. doi: 10.1053/j.gastro.2007.11.010. Epub 2007 Nov 12. PMID 18164296
- [Background] Everhart JE, Lok AS, Kim HY, Morgan TR, Lindsay KL, Chung RT, Bonkovsky HL, Ghany MG; HALT-C Trial Group. Weight-related effects on disease progression in the hepatitis C antiviral long-term treatment against cirrhosis trial. Gastroenterology. 2009 Aug;137(2):549-57. doi: 10.1053/j.gastro.2009.05.007. Epub 2009 May 13. PMID 19445938
- [Background] Romero-Gomez M, Del Mar Viloria M, Andrade RJ, Salmeron J, Diago M, Fernandez-Rodriguez CM, Corpas R, Cruz M, Grande L, Vazquez L, Munoz-De-Rueda P, Lopez-Serrano P, Gila A, Gutierrez ML, Perez C, Ruiz-Extremera A, Suarez E, Castillo J. Insulin resistance impairs sustained response rate to peginterferon plus ribavirin in chronic hepatitis C patients. Gastroenterology. 2005 Mar;128(3):636-41. doi: 10.1053/j.gastro.2004.12.049. PMID 15765399
- [Background] Mathias RA, Deepa M, Deepa R, Wilson AF, Mohan V. Heritability of quantitative traits associated with type 2 diabetes mellitus in large multiplex families from South India. Metabolism. 2009 Oct;58(10):1439-45. doi: 10.1016/j.metabol.2009.04.041. Epub 2009 Jul 1. PMID 19570552
- [Background] Arase Y, Suzuki F, Suzuki Y, Akuta N, Kobayashi M, Kawamura Y, Yatsuji H, Sezaki H, Hosaka T, Hirakawa M, Ikeda K, Kumada H. Sustained virological response reduces incidence of onset of type 2 diabetes in chronic hepatitis C. Hepatology. 2009 Mar;49(3):739-44. doi: 10.1002/hep.22703. PMID 19127513
- [Background] Idrees M, Riazuddin S. Frequency distribution of hepatitis C virus genotypes in different geographical regions of Pakistan and their possible routes of transmission. BMC Infect Dis. 2008 May 23;8:69. doi: 10.1186/1471-2334-8-69. PMID 18498666
- [Background] Peng JS, Wang X, Liu MQ, Zhou DJ, Gong J, Xu HM, Chen JP, Zhu HH, Zhou W, Ho WZ. Genetic variation of hepatitis C virus in a cohort of injection heroin users in Wuhan, China. Virus Res. 2008 Jul;135(1):191-6. doi: 10.1016/j.virusres.2008.01.017. Epub 2008 Mar 18. PMID 18353479
- [Background] Pearlman BL, Ehleben C, Saifee S. Treatment extension to 72 weeks of peginterferon and ribavirin in hepatitis c genotype 1-infected slow responders. Hepatology. 2007 Dec;46(6):1688-94. doi: 10.1002/hep.21919. PMID 18046717
- [Background] Sherman M, Shafran S, Burak K, Doucette K, Wong W, Girgrah N, Yoshida E, Renner E, Wong P, Deschenes M. Management of chronic hepatitis C: consensus guidelines. Can J Gastroenterol. 2007 Jun;21 Suppl C(Suppl C):25C-34C. PMID 17568824